CLINICAL TRIAL: NCT02165436
Title: The Use of Chewing Gum Reduces Post-operative Ileus and Gastrointestinal Complications in Pediatric Scoliosis Patients.
Brief Title: Chewing Gum Facilitates an Earlier Return to Bowel Function in Pediatric Scoliosis Patients: A Prospective Randomized Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Joseph G. Khoury, MD, Assistant Professor - Pediatric Orthopaedic Surgery, University of Alabama at Birmingham
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: X090615006
Record Dates: First submitted 2014-06-12; First posted 2014-06-17 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-06

CONDITIONS: Scoliosis
MeSH Terms: conditions — Scoliosis | interventions — Chewing Gum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): No gum
  Interventions: Other: Control
- Chewing Gum (Active Comparator): Bubble gum-flavored sugar-free gum - chew for 15-30 minutes 5 times/day
  Interventions: Other: Chewing gum

INTERVENTIONS:
Other: Chewing gum — Subjective assessment - subjective assessment of abdominal pain and nausea.
  Arms: Chewing Gum
Other: Control — No intervention will be assessed for this group.
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate the effectiveness of chewing gum on reducing post-operative ileus and reducing post-operative gastrointestinal symptoms in pediatric patients undergoing surgical correction of scoliosis. This study would provide minimal risk to its study population, and has the opportunity to provide a benefit to patients undergoing scoliosis surgery. If shown to be effective, this could lead to changes and improvement of the post-operative course for pediatric scoliosis patients.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise meets criteria for surgical correction of scoliosis
* Mental capacity to understand the purpose of the study
* Idiopathic scoliosis or neuromuscular scoliosis with mild cerebral involvement
* Posterior surgery approach only

Exclusion Criteria:

* Unable to safely chew gum due to oropharyngeal issues or airway issues
* History of GI surgery (G-tube, fundoplication, ostomy etc...)
* Anterior approach

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 83 (Actual)
Dates: Start 2009-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Time to return of normal bowel function. | 72-96 hours
  Patients are interviewed daily as inpatient and then several days after surgery to determine the time (reported in hours post-operative) first flatus and first bowel movement was experienced.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Khoury, MD, Principal Investigator — Pediatric Orthopaedic Surgery - University of Alabama At Birmingham
Locations (1):
- The Children's Hospital of Alabama, Birmingham, Alabama, United States